CLINICAL TRIAL: NCT04668027
Title: Evaluating the Efficacy of Impulse Oscillation Before and After Bronchial Provocation Test and Bronchial Dilation Test in Patients With Chronic Airway Disease
Brief Title: Impulse Oscillation to Evaluate Diagnostic Efficacy in Patients With Chronic Airway Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020LX0007_ZD
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Chronic Airway Disease
Keywords: impulse oscillation; bronchial provocation test; bronchial dilation test; asthma; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Bronchial Provocation Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chronic airway disease group (Experimental): Before the test, patients with FEV1/FVC≥0.7 are divided into the provocation test group, patients with FEV1/FVC <0.7 are divided into the dilation test group.
  Interventions: Diagnostic Test: impulse oscillation（IOS）; Diagnostic Test: bronchial provocation test(BPT); Diagnostic Test: bronchial dilation test(BDT)

INTERVENTIONS:
Diagnostic Test: impulse oscillation（IOS） — The patient is tested for the first IOS after the screening test, and performed the second IOS test immediately after the results of BPT or BDT. The patient takes seats, body relax, make sure the mouthpiece is fully covered by mouth, then clip nose with both hands to cover both sides of the cheek, and then calms breathing one minutes.
Diagnostic Test: bronchial provocation test(BPT) — Patient needs to cooperate with the inhalation of acetylcholine stimulants with low to high concentrations, and operates in accordance with the standard nebulized administration procedure. Measure FEV1 after each inhalation and take the high value. The interval between the inhalation of two adjacent doses is 5 minutes, until the FEV1 decrease value is ≥20% of the FEV1 base value or the highest inhalation concentration. The patient needs to cooperate to ensure that the filter is as tight as possible to prevent air leakage, and performs exhalation and inhalation with the greatest strength and fastest speed. After the examination,the patient should inhale the bronchodilator salbutamol sulfate (400ug).
Diagnostic Test: bronchial dilation test(BDT) — The patient inhales the salbutamol sulfate (400ug). 15 minutes later, the pulmonary function tester is used for measurement. The patient needs to cooperate to ensure that the filter is as tight as possible to prevent air leakage, and to exhale and breathe with the greatest strength and fastest speed. Inhale.

SUMMARY:
The aim of the research is to explore the diagnostic efficacy of impulse oscillation (IOS) before and after bronchial provocation test (BPT) and bronchial dilation test (BDT) in chronic airway disease.

DETAILED DESCRIPTION:
The present study has the following objectives:

to explore the diagnostic value of IOS before and after BPT/BDT in chronic airway disease, to assess the diagnostic accuracy of IOS in chronic airway disease with special regard to its discriminating value between asthma and chronic obstructive pulmonary disease, to evaluate the characteristics of airway resistance after BPT/BDT, to evaluate the airway reversibility and hyperresponsiveness（AHR）in asthma.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old, no gender limit;
2. The subject voluntarily cooperated with the research and signed an informed consent form;
3. Meet any of the following three criteria:

   * Patients with asthma, the standard diagnosis of asthma complied with the GINA 2019; ② Patients with COPD, the standard diagnosis of COPD complied with GOLD 2019; ③ The subjects in the healthy control group had normal vital capacity (baseline FEV1≥80% of the predicted value, FEV1/FVC was greater than the Lower Limit of Normal, and with negative result of BPT or BDT).

Exclusion Criteria:

1. History of other lung diseases, such as cystic fibrosis, bronchiolitis obliterans, tuberculosis, lung cancer, etc.;
2. After taking corticosteroid therapy in the last 4 weeks, respiratory tract infection occurred within 8 weeks;
3. A history of myocardial infarction and stroke in the past 3 months; a history of severe arrhythmia, severe cardiac insufficiency, and unstable angina in the past 4 weeks, etc.;
4. In the past 4 weeks, severe hemoptysis and epileptic seizures require medication; severe hyperthyroidism;
5. Pregnant women;
6. Other researchers consider it inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
The Value of the Change of IOS after BPT/BDT. | at least 4 weeks of treatment
  The value of respiratory reactance and resistance will be measured by Jaeger MasterScreen pulmonary function meter. And the main indicators that will be recorded are ΔZ5%、ΔR5%、ΔR20%、ΔR5-R20%、ΔR5-R20/R5%、ΔX5%、ΔAx% and ΔFres%. The receiver operating characteristic (Receiver Operating Characteristic, ROC) curve will be used to analyze the predictive value of IOS parameters for the positive results of BPT and BDT.
The Value of the Change of spirometry after BPT/BDT. | at least 4 weeks of treatment
  The value of spirometry will be performed with a spirometer (Jaeger, Hoechberg, Germany) in accordance with the specifications and performance criteria recommended in the American Thoracic Society (ATS)/European Respiratory Society (ERS) Standardization of Spirometry.And the main indicators that will be recorded are ΔFVC%、ΔFEV1%、ΔFEV1/FVC%、ΔMMEF%、ΔMEF75%、ΔMEF50% and ΔMEF25%.

CONTACTS AND LOCATIONS:
Overall Officials: Huapeng Yu, Principal Investigator — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No